CLINICAL TRIAL: NCT05193110
Title: Evaluation of CAD/CAM Versus Injection Molding Techniques of Polyetheretherketone (PEEK) Sub-periosteal Implant Retaining Maxillary Fixed Prosthesis
Brief Title: Two Years Follow up of Polyetheretherketone (PEEK) Sub-periosteal Implant Retaining Maxillary Fixed Prosthesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: A09091019
Record Dates: First submitted 2021-12-30; First posted 2022-01-14 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2021-12

CONDITIONS: Mastication Disorder
Keywords: Sub-periosteal implant; PEEK; CAD/CAM prosthesis; Maxilla
MeSH Terms: interventions — polyetheretherketone

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAD/CAM PEEK sub-periosteal implant retaining maxillary fixed prosthesis (Other): 4 PEEK sub-periosteal implants were surgically placed for patients demonstrated sever bone loss especially in the posterior region which complicate conventional implant placement for full arch prosthesis.The PEEK framework was fabricated by CAD/CAM method
  Interventions: Other: Polyetheretherketone (PEEK) Sub-periosteal Implant Retaining Maxillary Fixed Prosthesis
- Injection molding PEEK sub-periosteal implant retaining maxillary fixed prosthesis (Other): 4 CAD/CAM PEEK sub-periosteal implants were surgically placed for patients demonstrated sever bone loss especially in the posterior region which complicate conventional implant placement for full arch prosthesis.The PEEK framework was fabricated by injection molding technique method.
  Interventions: Other: Polyetheretherketone (PEEK) Sub-periosteal Implant Retaining Maxillary Fixed Prosthesis

INTERVENTIONS:
Other: Polyetheretherketone (PEEK) Sub-periosteal Implant Retaining Maxillary Fixed Prosthesis — Sub-periosteal Implant Retaining Maxillary Fixed Prosthesis fabricated by digital & milling technology

SUMMARY:
This clinical trial demonstrates prosthetic management of patients complained from lack of satisfaction and function of maxillary conventional complete denture as a result of severe maxillary ridge resorption seeking for fixed restoration. They were attended to the Department of Prosthodontics, Faculty of Dentistry, Mansoura University (Mansoura, Egypt). They demonstrated sever bone loss especially in the posterior region which complicate conventional implant placement for full arch prosthesis. Eight PEEK sub-periosteal implants were surgically placed. Probing depth was measured after three & six months from sub-periosteal implant placement. Tumor necrosis factor-alpha (TNF-α) & Interleukin-8(IL-8) Peri-abutment cervicular fluid were measured one month, three months , six months & one year from sub-periosteal implant placement. Clinical & Radiographic examination (CBCT) was done two years after sub-periosteal implant placement.

DETAILED DESCRIPTION:
Panoramic radiograph was done for each patient for diagnostic criteria, to evaluate condition of the ridge and to be a base line for further radiographic follow up examination . Fabrication of sub-periosteal implant was done as following: Computed tomography (CT) was done for each patient while wearing the denture with radio opaque markers and saved as STL file .CBCT was done for each denture and saved as STL file. Both STL files were aligned together to obtain a complete virtual model of the patient with all information about bone, soft tissue and the new prosthesis. This STL file then was processed and printed, in resin, using powerful rapid prototyping machine. The sub-periosteal implant was designed virtually on the virtual model by using dental wings(coDiagnostiXTM programme) .Location of the 4 abutments were designed to be on the canines and first molar region. Screws location were designed to be on compact bone, anterior nasal spine, hard palate and zygomatic bone .Height of the abutments were 5-6 mm..Thickness of the PEEK was 1.5 mm during construction and after finishing and polishing become 1.2 mm The sub-periosteal implant was then saved as an STL file, this file was first printed in resin to verify the accuracy of the fit on the 3D printed model of the patient . Finishing and polishing was done by PEEK polishing sets then the framework was decontaminated and packaged for sterilization by autoclave.

The surgery was done by a surgeon under local anaesthesia 4% Articaine with 1:100,000 epinephrine for hemostasis (articaine, Insiba, Spain) to the maxillary arch.The flap was done using three incision lines. the crestal incision was performed at the crest of the ridge, Two oblique releasing incisions were done at the distal ends of the crestal incision. Elevating the flap was done by the mucoperiosteal elevator. Sub-periosteal PEEK implant was placed and checked for its correct position, after placing the sub-periosteal implant, Fixation was done by 2mm diameter Fixation screws(AntonHipp,Germany) to the peek framework and bone. Continuous irrigation was done during drilling to avoid heat generation and bone necrosis. The flap was closed while the 4 abutments projecting from the flap using 3/0 resorbable vicryl sutures .1gm Amoxicillin was prescribed twice daily for every patient.Diclofenac potassium was prescribed to relieve pain.Chlorohexidine mouth wash was prescribed to decrease inflammation and swelling. Instruction was given to both patients for soft diet for 1 weak, cold fomentations and not to move the check muscle strongly to avoid releasing of the sutures. Patients were instructed to periodic recall every 2 week for 6 weeks. The implant was left for healing then evaluation of soft probing depth around the abutments were done three months & six months after surgical placement. For all surfaces Buccal(B), Palatal(P), Mesial(M), Distal(D). (TNF-α) & (IL-8) Peri-abutment cervicular fluid was detected by paper points & transferred to laboratory, specimens were evaluated by ELISA test one month ,three months , six months & 12 months after surgical placement. Clinical & Radiographic (CBCT) examination was done after 2 years from sub-periosteal implant placement.

After complete healing of the soft tissue, preparation was done to the PEEK abutments under copious irrigation with saline to avoid heat generation. Finishing and polishing of the PEEK abutments were done by using composite polishing instruments. Impression was taken to the maxillary arch using addition silicon impression material (Heavy and light body) in one step. Proper vertical dimension was recorded, and then Face-bow transfer record was done to orient the maxillary cast to the semi-adjustable articulator. Horizontal jaw relation was recorded; centric inter-occlusal record was made. The mandibular denture was mounted on the articulator using centric inter-occlusal wax record. PEEK framework was done for the abutments; Setting up all the artificial teeth was made on the articulator. The maxillary PEEK framework with teeth were tried in the patient's mouth then processed in to final prosthesis .Temporary cement was used after insertion of the prosthesis to enable peri-implant probing depth & cerivicular fluid evaluation then final cementation of the fixed prosthesis was done by DTK. Strict oral hygiene measures & electric water jet irrigator tooth brush was instructed for each patient

ELIGIBILITY:
Inclusion Criteria:• No systemic diseases or local pathosis that may affect bone healing. This will be verified through medical history, laboratory investigation and clinical examination by the physician.

* Completely edentulous maxillary and mandibular arch..
* Residual ridge covered by sufficient thickness of mucosa 2-3 mm as verified by probing depth by using plastic probe.
* All patients with maxillary insufficient bone quantity (horizontal and vertical dimensions) and insufficient bone quality D5(Housefields Units <) making it impossible to place root-form dental implants with a diameter of at least 3 mm and a length of at least 8 mm .as verified by CT.
* Sufficient inter-arch space as verified by probing.
* sufficient restorative space as verified by putty index technique
* Patient seeking for fixed prosthesis

Exclusion Criteria:

* Patients with absolute contraindications for surgical procedures such as: active cancer ,immunocompromised patients
* Patients with relative contraindications such as: patients with history of para functional habits (bruxism, clenching), bad habits as heavy smoking and alcoholism.. Also patients with history of radiation therapy in the head and neck region
* Patients with contraindication for grafting procedures.
* Non cooperative patients neither who don't attend regular appointments nor following the instructions during construction procedures

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-12-23 (Actual); Primary Completion 2021-12-02 (Actual); Study Completion 2021-12-28 (Actual)

PRIMARY OUTCOMES:
Polyetheretherketone (PEEK) Sub-periosteal Implant Retaining Maxillary Fixed Prosthesis. | 1 year
  PEEK sub-periosteal implants were surgically placed. Probing depth was measured after three & six months from sub-periosteal implant placement. Tumor necrosis factor-alpha (TNF-α) & Interleukin-8(IL-8) Peri-abutment cervicular fluid were measured one month, three months , six months & one year from sub-periosteal implant placement.

CONTACTS AND LOCATIONS:
Overall Officials: Salah A. Hegazy, PhD, Study Chair — salahhegazy2003@yahoo.com
Locations (1):
- Faculty of dentistry , Mansoura University, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No